CLINICAL TRIAL: NCT03562403
Title: Deep Brain Stimulation in the Treatment of Intractable Movement Disorders ( Parkinson's Disease, Essential Tremors and Dystonia)
Brief Title: DBS in the Treatment of Intractable Movement Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Radwan Nouby, Assistant Lecturer in the Department of Neurosurgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS in movement disorders
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease, Essential Tremors and Dystonia
Keywords: deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS on patients with abnormal movement disorders (Experimental): 16 patients with intractable abnormal movement disorders (Parkinson's disease, Essential tremors and Dystonia)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — stimulation of different basal ganglionic nuclei by a inserting a device

SUMMARY:
The aim of this study is to observe the efficacy of Deep Brain Stimulation in the treatment of Parkinson's disease,Essential Tremors and Dystonia in our locality.

DETAILED DESCRIPTION:
Movement disorders are clinical syndromes result from disturbances of basal ganglia function with either an excess of movement or a paucity of voluntary and involuntary movements, unrelated to weakness or spasticity. Movement disorders are synonymous with basal ganglia or extrapyramidal diseases. Movement disorders are conventionally divided into two major categories-hyperkinetic and hypokinetic.

Hyperkinetic movement disorders refer to excessive, often repetitive, involuntary movements that intrude upon the normal flow of motor activity and it includes include Essential Tremors, Dystonia, Chorea, Dyskinesia, and Athetosis.

Hypokinetic movement disorders refer to akinesia (lack of movement), hypokinesia (reduced amplitude of movements), bradykinesia (slow movement) and rigidity. In primary movement disorders, the abnormal movement is the primary manifestation of the disorder. In secondary movement disorders, the abnormal movement is a manifestation of another systemic or neurological disorder.

The basal ganglia include the striatum (caudate. putamen, nucleus accumbens), the subthalamic nucleus (STN), the globuspallidus [internal segment. external segment, ventral pallidum (VP)]. and the substantianigra pars compacta (SNpc) and substantianigra pars reticulata (SNpr).

Surgical therapies for the treatment of movement disorders can be divided into two broad categories: ablative and restorative. The most common structures targeted during stereotactic surgery for movement disorders are the motor thalamus, the globuspallidus internus and the subthalamic nucleus. Ablative surgical therapies for Movement disorders include thalamotomy and pallidotomy. Restorative surgical therapies include deep brain stimulation and transplantation of fetal tissue, cell lines that express trophic factors, or somatically delivered gene therapies. The theoretical advantage of Deep Brain Stimulation over ablative procedures is the lack of tissue destruction especially with deep brain stimulation. This is particularly appealing for patients needing bilateral procedures.

Parkinson's disease is the best example of a hypokinetic movement disorder. The interest in surgery has been prompted by the growing realization of the limitations of drug therapy for these movement disorders, improvement in neuroimaging capabilities, enhanced stereotactic surgical techniques and better understanding of functional organization of the basal ganglia and its pathophysiology of these movement disorders. There are many theories on how does Deep Brain Stimulation works in the treatment of movement disorders, these theories include Neurostimulation, Neuroinhibition, and Release of neurotransmitters. Deep brain has the following advantages over ablative surgery: No destruction of brain tissue can adjust stimulus parameters, Perform bilateral operations, significant reduction (50-75%) in medication, and it is completely reversible.

Since the introduction of deep brain stimulation almost 20 years ago, there has been an immense resurgence in interest in the surgical technique. However, the investigators are still asking some of the same questions. How can the investigators improve the targeting? What is the optimal target? In addition, the investigators have started asking some new questions such as how does deep brain stimulation work, and what other disorders can deep brain stimulation be applied to?

ELIGIBILITY:
Inclusion Criteria:

1. Dopa responsiveness
2. Minimum disease duration of 5 years.
3. Diagnosis of idiopathic Parkinsons disease
4. Patients with intractable Essential Tremors.
5. Patients with intractable dystonia

Exclusion Criteria:

1. Significant medical health problems.
2. Significant cognitive impairment
3. Bleeding tendencies

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in the unified parkinson's disease rating scale score | baseline(pre-DBS )and 6 months post-DBS
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a commonly used survey tool used to assess symptom severity of patients with Parkinson's disease (PD). It covers several different domains including 1) thought, behavior and mood 2) activities of daily living 3) motor activity 4) complications of therapy and others.
  Part I: evaluation of mentation, behavior, and mood Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food Part III: clinician-scored monitored motor evaluation Part IV: complications of therapy Part V: Hoehn and Yahr staging of severity of Parkinson's disease Part VI: Schwab and England ADL scale

SECONDARY OUTCOMES:
Change in antiparkinsonian medication use | baseline(pre-DBS and 6 months post-DBS
  the percent in reduction of antiparkinsonian medications used after DBS

CONTACTS AND LOCATIONS:
Overall Officials: Amr Elnaggar, MD, Study Director — University of Louisville

REFERENCES:
- [Result] Guttman M, Kish SJ, Furukawa Y. Current concepts in the diagnosis and management of Parkinson's disease. CMAJ. 2003 Feb 4;168(3):293-301. PMID 12566335
- [Result] Jankovic J, Cardoso F, Grossman RG, Hamilton WJ. Outcome after stereotactic thalamotomy for parkinsonian, essential, and other types of tremor. Neurosurgery. 1995 Oct;37(4):680-6; discussion 686-7. doi: 10.1227/00006123-199510000-00011. PMID 8559296